CLINICAL TRIAL: NCT00581568
Title: Cutaneous Effects of Cryogen Spray Cooling
Acronym: CSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Wangcun Jia, PhD., Research Scientist, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20033200
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pain
Keywords: Skin cooling during laser treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Effects of Cryogen Spray Cooling (Experimental): Cutaneous Effects of Cryogen Spray Cooling
  Interventions: Other: Cutaneous Effects of Cryogen Spray Cooling

INTERVENTIONS:
Other: Cutaneous Effects of Cryogen Spray Cooling — Cutaneous Effects of Cryogen Spray Cooling
  Other Names: CSC

SUMMARY:
Cryogen Spray Cooling spurt is applied to the skin surface immediately before laser exposure. As liquid cryogen rapidly evaporates, the superficial skin temperature is reduced as a result of supplying the latent heat of vaporization. Tetrafluoroethane, an environmentally compatible, non-toxic, non-flammable freon substitute, has been demonstrated in multiple studies to be a safe and effective cooling agent and is the only cryogenic compound currently approved for dermatologic use by the Food and Drug Administration.

DETAILED DESCRIPTION:
The researcher can use laser treatment in combination with Cryogen Spray Cooling. The specific aim of this study is to characterize the clinical cutaneous effects of varying spurt durations and spurt delivery patterns that spurt durations of 100 ms or less will result in a very low incidence (less than 2%) of clinical skin effects (redness, blistering, local skin allergic reaction or skin discoloration) in any skin type.

Researchers can use Cryogen Spray Cooling to protect the skin epidermis during laser therapy to decrease treatment pain, allow safe treatment of darker skin types, and safe use of high laser fluences. Cryogen Spray Cooling with Tetrafluoroethane has been incorporated into many Food and Drug Administration approved, commercially available laser devices currently used for treatment of vascular lesions, hair removal and non-ablative skin rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older

Exclusion Criteria:

* Age <18
* History of cold sensitivity
* Inflammatory rash on the test site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Skin cooling during laser treatment | 1 minute
  Cryogen Spray Cooling spray cooling skin during laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D.,Ph.D, Study Chair — Beckman Laser Institute; Wangcun Jia, PhD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute Medical and Surgical clinic, Irvine, California, United States